CLINICAL TRIAL: NCT06772038
Title: Dynamic Assessment of Fluid Responsiveness and Venous Congestion: Evolution of the VExUS Score During Volume Expansion
Brief Title: Fluid Responsiveness and Venous Congestion Evolution During Volume Expansion
Acronym: FREVO
Status: Recruiting | Type: Observational
Sponsor: Bicetre Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Longgang District People's Hospital of Shenzhen (Other)
Responsible Party: Principal Investigator, Xavier Monnet, Professor Xavier Monnet, MD, PHD, Bicetre Hospital
Other Study IDs: 2022-A00580-43
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Hemodynamic; Fluid Responsiveness; Venous Congestion; Fluid Challenge
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fluid Responder: Patients with an aumentation of cardiac index>= 15% after a fluid challenge
- Fluid Non-responder: Patients without an aumentation of cardiac index>= 15% after a fluid challenge

SUMMARY:
Fluid responsiveness is a critical determinant guiding fluid therapy in critically ill patients. However, excessive fluid administration can result in fluid overload, leading to venous congestion and worse clinical outcomes. Venous congestion, a marker of impaired fluid clearance, is increasingly recognized as a significant contributor to poor prognosis. Previous studies have demonstrated the coexistence of fluid responsiveness and venous congestion in critically ill patients. Notably, these studies were limited by the absence of fluid challenge-the gold standard for assessing fluid responsiveness-leaving the dynamic relationship between fluid responsiveness and venous congestion incompletely understood. This study aims to investigate the interplay and temporal evolution of fluid responsiveness and venous congestion following a standardized fluid challenge in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized in the intensive care unit (ICU)
* Hemodynamic monitoring in place, with a pulse wave contour analysis- derived estimation of cardiac output (either calibrated or uncalibrated)
* Decision made by clinicians to perform volume expansion through intravenous infusion of crystalloid fluid

Exclusion Criteria:

* Pregnancy
* Refusal to participate by relatives of the patient or the patient himself

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with evidence of inadequate tissue perfusion, who are already monitored using a pulse wave contour analysis-derived estimation of cardiac output (either calibrated or uncalibrated)，and for whom clinicians have decided to administer volume expansion through intravenous crystalloid infusion.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
The difference in venous congestion (VExUS) changes between fluid responders and non-responders following a fluid challenge. | before and after 15-minute fluid challenge.

SECONDARY OUTCOMES:
The differential evolution of venous congestion (VExUS) changes between fluid responders and non-responders 1 hour after a fluid challenge. | 1 hour after fluid challenge

CONTACTS AND LOCATIONS:
Locations (3):
- China (2):
  - First affiliated Hospital , Sun Yat-sen University, Guangzhou, Guangdong
  - Longgang Central Hospital of Shenzhen, Shenzhen, Guangdong
- Bicetre Hospital, Paris, Val-de-Marne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Munoz F, Born P, Bruna M, Ulloa R, Gonzalez C, Philp V, Mondaca R, Blanco JP, Valenzuela ED, Retamal J, Miralles F, Wendel-Garcia PD, Ospina-Tascon GA, Castro R, Rola P, Bakker J, Hernandez G, Kattan E. Coexistence of a fluid responsive state and venous congestion signals in critically ill patients: a multicenter observational proof-of-concept study. Crit Care. 2024 Feb 19;28(1):52. doi: 10.1186/s13054-024-04834-1. PMID 38374167
- [Background] Monnet X, Shi R, Teboul JL. Prediction of fluid responsiveness. What's new? Ann Intensive Care. 2022 May 28;12(1):46. doi: 10.1186/s13613-022-01022-8. PMID 35633423
- [Background] Messina A, Calabro L, Pugliese L, Lulja A, Sopuch A, Rosalba D, Morenghi E, Hernandez G, Monnet X, Cecconi M. Fluid challenge in critically ill patients receiving haemodynamic monitoring: a systematic review and comparison of two decades. Crit Care. 2022 Jun 21;26(1):186. doi: 10.1186/s13054-022-04056-3. PMID 35729632
- [Background] Monnet X, Malbrain MLNG, Pinsky MR. The prediction of fluid responsiveness. Intensive Care Med. 2023 Jan;49(1):83-86. doi: 10.1007/s00134-022-06900-0. Epub 2022 Nov 3. No abstract available. PMID 36323911
- [Background] Joseph A, Petit M, Vignon P, Vieillard-Baron A. Fluid responsiveness and venous congestion: unraveling the nuances of fluid status. Crit Care. 2024 Apr 26;28(1):140. doi: 10.1186/s13054-024-04930-2. No abstract available. PMID 38671461